CLINICAL TRIAL: NCT02675556
Title: A Phase I, Prospective, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Potential Efficacy of Allogeneic Human Mesenchymal Stem Cell Infusion Versus Placebo in Patients With Treatment Resistant Depression.
Brief Title: Allogeneic Human Mesenchymal Stem Cells (hMSCs) Infusion in Patients With Treatment Resistant Depression
Acronym: ANU
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty in recruitment and funding.
Sponsor: Joshua M Hare (Other)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Sponsor - Investigator, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20140917
Record Dates: First submitted 2016-02-01; First posted 2016-02-05 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Treatment Resistant Depression
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Allogeneic hMSCs (Experimental): Forty (40) subjects will be treated with a single administration of allogeneic Human Mesenchymal Stem Cell (hMSCs): 100 x 10^6 (100 million) allo-hMSCs of cells delivered via a single peripheral intravenous infusion.
  Interventions: Drug: Allo-hMSCs
- Placebo (Placebo Comparator): Forty (40) subjects will be treated with a placebo administration consisting of 1% human albumin serum in Plasma-Lyte A delivered via a single peripheral intravenous infusion.
  Interventions: Drug: Placebo
- Pilot - Allogeneic hMSCs (Experimental): Eight (8) subjects will be treated with a single administration of allogeneic Human Mesenchymal Stem Cell (hMSCs): 100 x 10^6 (100 million) allo-hMSCs of cells delivered via a single peripheral intravenous infusion.
  Interventions: Drug: Allo-hMSCs

INTERVENTIONS:
Drug: Allo-hMSCs — a single administration of allogeneic Human Mesenchymal Stem Cell (hMSCs): 100 x 10^6 (100 million) allo-hMSCs of cells
  Other Names: Allogeneic Human Mesenchymal Stem Cells; Stem Cells
  Arms: Allogeneic hMSCs; Pilot - Allogeneic hMSCs
Drug: Placebo — a placebo administration consisting of 1% human albumin serum in Plasma-Lyte A
  Arms: Placebo

SUMMARY:
This study is intended to evaluate the safety and potential efficacy of Allogeneic Human Mesenchymal Stem Cell Infusion versus placebo in patients with Treatment Resistant Depression.

DETAILED DESCRIPTION:
This is a phase I study, with eight subjects in the pilot phase and eighty (80) subjects fulfilling all inclusion/exclusion criteria's will be randomly assigned to receive allogeneic Human Mesenchymal Stem Cell (hMSCs) or placebo in a 1:1 blinded fashion.

The 8 subjects in the pilot phase will receive a single infusion of 100 million hMSCs.

40 patients will receive a single administration of allogeneic hMSCs and another 40 patients will receive a single administration of Placebo in a 1:1 blinded fashion.

Following infusion, patients will be followed at 2, 4, 6, 8, 10 and 12 week's post-infusion to complete all safety and efficacy assessments. During these 12 weeks starting after the week 2 visit subjects will have a phone call in-between their visits. Patients will additionally be followed for up to 12 months post-infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Subjects age equal or greater than 18 and equal or less than 75 years at the time of signing the Informed Consent Form.
3. Diagnosis of Treatment resistant depression (Failed at least two adequate trials of antidepressant monotherapy or antidepressant augmentation with an antipsychotic or lithium during the current episode)
4. Patients who are receiving a third or more treatment will only be entered if they have not responded to the current treatment.
5. Experiencing a current Major Depressive Episode (fulfilling Structured clinical interview for Diagnostic and Statistical Manual of Mental Disorders (DSM V) criteria per Structured Clinical Interview for DSM (SCID) for categorical diagnosis, and the Hamilton Depression Rating Scale for Depression (HAM-D))
6. Hamilton Depression Rating Scale 21-item score greater than 18
7. Adequacy of previous failed antidepressant trials will be defined using standard criteria by Massachusetts General Hospital (MGH) of patients with a score greater than or equal to 2.5
8. Increased inflammation ([Serum CRP] greater than 3.0 mg/L)

Exclusion Criteria:

In order to participate in this study, a patient Must Not:

1. Women who are pregnant, nursing, or of childbearing potential, while not practicing effective contraceptive methods. (Female subjects of childbearing potential must undergo a serum or urine pregnancy test at screening and within 36 hours prior to infusion.)
2. Inability to perform any of the assessments required.
3. Have clinically significant abnormal screening laboratory values, including but not limited to: hemoglobin <8 g/dl, white blood cell count <3000/mm3, platelets<80,000/mm3, INR > 1.5 not due to a reversible cause (i.e. Coumadin), aspartate transaminase, alanine transaminase, or alkaline phosphatase > 3 times upper limit of normal, total bilirubin > 1.8 mg/dl (unless due to a benign cause).
4. Active medical condition that could cause or exacerbate depressive symptoms (e.g., hypothyroidism, anemia)
5. Serious comorbid illness or any other condition (Such as bipolar, schizophrenia or schizoaffective disorder) that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study.
6. Have acute suicidality
7. Prior history of a suicide attempt, within the past year.
8. Active psychotic disorder, eating disorder, or substance use disorder within 6 months of enrollment
9. Treatment with any medication that, in the opinion of the Investigator, may compromise the safety of the subject or affect the validity of the data or the study endpoints.
10. First major depressive episode after 50 years of age.
11. Have known allergies to penicillin or streptomycin.
12. Have hypersensitivity to dimethyl sulfoxide (DMSO).
13. Have a clinical history of malignancy within 5 years (i.e., subjects with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ or cervical carcinoma.
14. Have a non-pulmonary condition that limits lifespan to < 1 year.
15. Have a history of drug or alcohol abuse within the past 24 months.
16. Be serum positive for HIV, hepatitis BsAg or Viremic hepatitis C.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of any treatment-emergent serious adverse events (TE-SAEs) | One month post infusion
  defined as a composite of acute suicidality, and hospitalization for suicide attempts.

SECONDARY OUTCOMES:
Reduction of Inflammation | Week 12
  Reduction of Inflammation: Change in serum concentrations of high sensitivity C-Reactive Protein (hs-CRP)

OTHER OUTCOMES:
Reductions in serum concentrations | Week 12
  Reductions in serum concentrations of other inflammatory markers;
Reduction in Depressive Symptoms | Week 12
  Reduction in Depressive Symptoms due to change in Montgomery-Asberg Depression Rating Scale (MADRS)
Reduction in Anhedonia | Week 12
  Reduction in Anhedonia due to change in the Snaith Hamilton Pleasure Scale
Improvements in Cognition | Week 12
  Improvements in Cognition as a result of changes in Brief Assessment of Cognition for Affective Disorders (BAC-A), Performance Based Skills Assessment (UPSA-B), and Specific Level of Functioning (SLOF) scores
Improvements in Functional Capacity | Week 12
  Improvements in Functional Capacity as a result of changes in Brief Assessment of Cognition for Affective Disorders (BAC-A), Performance Based Skills Assessment (UPSA-B), and Specific Level of Functioning (SLOF) scores
Improvements in everyday functioning | Week 12
  Improvements in everyday functioning as a result of changes in Brief Assessment of Cognition for Affective Disorders (BAC-A), Performance Based Skills Assessment (UPSA-B), and Specific Level of Functioning (SLOF) scores
Mediating effects of child abuse and neglect. | week 12
  Mediating effects of child abuse and neglect.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Hare, MD, Study Director — ISCI / University of Miami Miller School of Medicine
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided